CLINICAL TRIAL: NCT06493409
Title: A Phase I, Two-part, Single-center, Open-label, Drug-drug Interaction Study to Assess the Effect of Voriconazole (Part 1) and Quinidine (Part 2) on the Pharmacokinetics of a Single Dose of Repotrectinib (BMS-986472) in Healthy Participants
Brief Title: A Study to Assess the Effect of Voriconazole and Quinidine on the Pharmacokinetics of a Single Dose of Repotrectinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA127-1072
Expanded Access: NCT05926232 (Available)
Record Dates: First submitted 2024-06-25; First posted 2024-07-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: drug interaction; healthy; repotrectinib; BMS-986472; pharmacokinetics
MeSH Terms: interventions — repotrectinib; Voriconazole; Quinidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental)
  Interventions: Drug: Repotrectinib; Drug: Voriconazole
- Part 2 (Experimental)
  Interventions: Drug: Repotrectinib; Drug: Quinidine

INTERVENTIONS:
Drug: Repotrectinib — Specified dose on specified days
  Other Names: BMS-986472
Drug: Voriconazole — Specified dose on specified days
  Arms: Part 1
Drug: Quinidine — Specified dose on specified days
  Arms: Part 2

SUMMARY:
The purpose of this study is to evaluate the effects of coadministration of voriconazole or quinidine on the pharmacokinetics (PK) of repotrectinib in healthy male and female (individual not of childbearing potential [INOCBP]) participants.

ELIGIBILITY:
Inclusion Criteria

* Healthy male and female individual(s) not of childbearing potential (INOCBP) participants of any race or ethnicity, as determined by no clinically significant findings in medical history, physical examination, 12-lead ECG, or vital signs as determined by the investigator or designee.
* Potassium, magnesium, and calcium at or above the lower limit of normal. For other clinical laboratory parameters, no clinically significant findings as determined by the investigator or designee.
* Must have a body mass index between 18 and 30 kg/m2 (inclusive) and body weight ≥ 50 kg at the time of signing the ICF.

Exclusion Criteria

* History of clinically significant acute or chronic medical illness, such as endocrine, gastrointestinal (GI), cardiovascular, peripheral vascular, hematological, hepatic, immunological, renal, respiratory, neoplastic, or genitourinary abnormalities/diseases as determined by the investigator or designee.
* History of GI disease or surgery that could possibly affect drug absorption, distribution, metabolism, and excretion (ADME) (eg, bariatric procedure, cholecystectomy). Uncomplicated appendectomy and hernia repair are acceptable.
* Gilbert's syndrome.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 23
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to Day 23
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to Day 23

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to Day 52
Number of participants with Severe Adverse Events (SAEs) | Up to Day 52
Number of participants with physical examination abnormalities | Up to Day 23
Number of participants with vital sign abnormalities | Up to Day 23
Number of participants with electrocardiogram abnormalities | Up to Day 23
Number of participants with clinical safety laboratory test abnormalities | Up to Day 22
Time of maximum observed plasma concentration (Tmax) | Up to Day 23
Apparent terminal phase half-life (T-HALF) | Up to Day 23
Apparent total body clearance (CLT/F) | Up to Day 23
Apparent volume of distribution of terminal phase (Vz/F) | Up to Day 23
Cmax | Up to Day 23
Area under the plasma concentration-time curve over one dosing interval (AUC(TAU)) | Up to Day 23
Trough observed plasma concentration (Ctrough) | Up to Day 23

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Fortrea - Daytona Beach, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com